CLINICAL TRIAL: NCT01795651
Title: Identification of Take Home Message in Lecture Based Learning: a Randomize Controlled Trial
Brief Title: Identification of Take Home Message in Lecture Based Learning
Acronym: T-REX 2
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0143
Record Dates: First submitted 2013-02-04; First posted 2013-02-21 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Educational Modules Given to French Juniors Taking the Postgraduate Critical Care Diploma
Keywords: teaching; knowledge translation; ICU; postgraduate; lecture

GROUPS / COHORTS (1):
- Take-Home message
  Interventions: Procedure: identification of take-home message of lecture

INTERVENTIONS:
Procedure: identification of take-home message of lecture

SUMMARY:
Medical education involves the acquisition of a large quantity of information. Lecture-based learning (LBL) is the best known of conventional teaching methods. Two thirds of critical care junior doctors identified at best only one of the three main take-home messages of a lecture, suggesting that knowledge transfer is poor during passive format learning.

The investigators assess the impact of an intervention including the identification of take-home message of lecture with slides calling "Learning Objectives", "Message", "Conclusion", in the identification of take-home message in critical care junior doctors.

DETAILED DESCRIPTION:
Medical education involves the acquisition of a large quantity of information. Lecture-based learning (LBL) is the best known of conventional teaching methods. The main purpose of a lecture is knowledge transfer [1] and its great advantage is that of transferring knowledge from one individual to several or many. Knowledge transfer via LBL is still widely used in international medical congresses, in continuing medical education online via downloading of lectures offered by leading medical schools, and in postgraduate medical education in several countries. We showed that in prospective study of 13 lectures that two thirds of critical care junior doctors identified at best only one of the three main take-home messages of a lecture, suggesting that knowledge transfer is poor during passive format learning.

In this study, we assess the impact of an intervention including the identification of take-home message of lecture with slides calling "Learning Objectives", "Message", "Conclusion", in the identification of take-home message in critical care junior doctors.

6 lectures are performed by professor without specific orders. 6 lectures are performed by professor with the intervention. Both groups of professors do not know this study The critical care juniors do not know the intervention. We compare the take-home messages of students with those of lecturer, 1 month after the lecture.

ELIGIBILITY:
Inclusion Criteria:

* critical care junior who attends lecture

Exclusion Criteria:

* refusal
* critical care junior who do not speak french

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French juniors
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of match lecturer's take home message | 1 month after the lecture

SECONDARY OUTCOMES:
Measure of correct responses to multiple choice-questions | 1 month after the lecture

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre LAUTRETTE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Lautrette A, Boyer A, Gruson D, Argaud L, Schwebel C, Tardy B, Vignon P, Megarbane B, Schoeffler P, Chabrot P, Schmidt J, Boirie Y, Guerin C, Darmon M, Klouche K, Souweine B, Dellamonica J, Pereira B; TREX group. Impact of take-home messages written into slide presentations delivered during lectures on the retention of messages and the residents' knowledge: a randomized controlled study. BMC Med Educ. 2020 Jun 3;20(1):180. doi: 10.1186/s12909-020-02092-7. PMID 32493318